CLINICAL TRIAL: NCT05614076
Title: Clinical Performance Of Conserved Chalky White Demineralized Enamel Cavity Margins Versus Totally Removed Carious Margins In Class V Cavities Restored With Composite Resin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maryam Salim Dawood, main investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422019474770
Record Dates: First submitted 2022-06-09; First posted 2022-11-14 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Class V Dental Caries

STUDY DESIGN:
Intervention Model Description: 1:1
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservation of the demineralized chalky white enamel margin of class V cavities (Experimental): for cavity design in this arm we Conserved the demineralized chalky white enamel margin of class V cavities then application of resin composite restoration
  Interventions: Procedure: conserved chalky white enamel margins of class V cavities
- Total removal of demineralized enamel margin of class V cavities (Active Comparator): for cavity design in this arm is Total removal of demineralized enamel margin of class V cavities and restoration with resin composite
  Interventions: Procedure: Total removal of demineralized enamel margins of class V cavities

INTERVENTIONS:
Procedure: conserved chalky white enamel margins of class V cavities — during cavity preparation, we conserved chalky white enamel margins of class V cavities and then restored them with resin composite restorations,we assessed the restorations with visual inspection using a mirror and explorer according to USPHS Criteria
  Arms: Conservation of the demineralized chalky white enamel margin of class V cavities
Procedure: Total removal of demineralized enamel margins of class V cavities — during cavity preparation, we removed the total chalky white enamel margins of class V cavities and then restored them with resin composite restorations, we assessed the restorations with visual inspection using a mirror and explorer according to USPHS Criteria
  Arms: Total removal of demineralized enamel margin of class V cavities

SUMMARY:
This study aims to compare the clinical performance of conserved chalky white demineralized enamel margins with total removal of demineralized enamel margins in class v cavities restored with composite in patients with acute carious cervical lesions

DETAILED DESCRIPTION:
With limited evidence-based information about the clinical performance of conserved white chalky enamel margins in class v .it is beneficial to compare the newly concept of preserved the white chalky deminerlized enamel margins using a randomized clinical trial to test the null hypothesis that this new concept has the same clinical performance as total removal of demineralized enamel margins in class v cavities restored with composite in patients with acute carious cervical lesions .The comparator will be the concept of total removal of demineralized enamel margins in class v cavities restored with composite Patients are selected according to the eligibility criteria, Local anesthesia will be administered and the operative field will be isolated before starting the restorative procedure. For the comparator group, standard class V cavities will be prepared at labial surface with totally removed carious enamel margins. For interventional group, class V cavity prepared at labial surface with preserved the chalky demineralized enamel margins then applications of remineralizing agent(MI paste plus) before the application of resin composite restoration. Local anesthesia will be administered and the operative field will be isolated before starting the restorative procedure. For control group, standard class V cavities will be prepared at labial surface with totally removed carious enamel margins. For experimental group, class V cavity prepared at labial surface with preserved the chalky demineralized enamel margins then applications of remineralizing agent(MI paste plus) before the application of resin composite restoration. both cavities groups restored with resin composite restorations. The restorations are assessed using the modified USPHS criteria at the time intervals stated in the outcome measures

ELIGIBILITY:
Inclusion Criteria:

* class V carious lesions in premolars and molars.
* Vital upper or lower teeth with no signs of irreversible pulpitis.
* Presence of favorable occlusion and teeth are in normal contact with the adjacent teeth.

Exclusion Criteria:

* Deep carious defects (close to pulp, less than 1 mm distance).
* Periapical pathology or signs of pulpal pathology.
* Endodontically treated teeth
* Tooth hypersensitivity.
* Possible prosthodontic restoration of teeth.
* Heavy occlusion or occlusal contacts or history of bruxism.
* Severe periodontal affection

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
marginal discoloration | 3 months
  ordinal criteria scoring system (ordinal)
marginal discoloration | 6 months
  ordinal criteria scoring system (ordinal)
marginal discoloration | 12 months
  ordinal criteria scoring system (ordinal)

SECONDARY OUTCOMES:
color change | 3 month
  ordinal criteria scoring system (ordinal)
color change | 6 month
  ordinal criteria scoring system (ordinal)
color change | 12 month
  ordinal criteria scoring system (ordinal)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdalla AI, Garcia-Godoy F. Clinical performance of a self-etch adhesive in Class V restorations made with and without acid etching. J Dent. 2007 Jul;35(7):558-63. doi: 10.1016/j.jdent.2007.02.006. Epub 2007 Apr 27. PMID 17467137
- [Background] Alexandria AK, Nassur C, Nobrega CBC, Valenca AMG, Rosalen PL, Maia LC. In situ effect of titanium tetrafluoride varnish on enamel demineralization. Braz Oral Res. 2017 Nov 6;31:e86. doi: 10.1590/1807-3107BOR-2017.vol31.0086. PMID 29116298
- [Background] Bayne SC, Schmalz G. Reprinting the classic article on USPHS evaluation methods for measuring the clinical research performance of restorative materials. Clin Oral Investig. 2005 Dec;9(4):209-14. doi: 10.1007/s00784-005-0017-0. No abstract available. PMID 16421996
- [Background] Baratieri LN, Ritter AV. Critical appraisal. To bevel or not in anterior composites. J Esthet Restor Dent. 2005;17(4):264-9. doi: 10.1111/j.1708-8240.2005.tb00126.x. PMID 16231497
- [Background] Chen H, Liu X, Dai J, Jiang Z, Guo T, Ding Y. Effect of remineralizing agents on white spot lesions after orthodontic treatment: a systematic review. Am J Orthod Dentofacial Orthop. 2013 Mar;143(3):376-382.e3. doi: 10.1016/j.ajodo.2012.10.013. PMID 23452972
- [Background] Kielbassa AM, Ulrich I, Schmidl R, Schuller C, Frank W, Werth VD. Resin infiltration of deproteinised natural occlusal subsurface lesions improves initial quality of fissure sealing. Int J Oral Sci. 2017 Jun;9(2):117-124. doi: 10.1038/ijos.2017.15. Epub 2017 Jun 16. PMID 28621326
- [Background] Korner P, El Gedaily M, Attin R, Wiedemeier DB, Attin T, Taubock TT. Margin Integrity of Conservative Composite Restorations after Resin Infiltration of Demineralized Enamel. J Adhes Dent. 2017;19(6):483-489. doi: 10.3290/j.jad.a39280. PMID 29152623
- [Background] Lata S, Varghese NO, Varughese JM. Remineralization potential of fluoride and amorphous calcium phosphate-casein phospho peptide on enamel lesions: An in vitro comparative evaluation. J Conserv Dent. 2010 Jan;13(1):42-6. doi: 10.4103/0972-0707.62634. PMID 20582219
- [Background] Koc Vural U, Kerimova L, Kiremitci A. Clinical comparison of a micro-hybride resin-based composite and resin modified glass ionomer in the treatment of cervical caries lesions: 36-month, split-mouth, randomized clinical trial. Odontology. 2021 Apr;109(2):376-384. doi: 10.1007/s10266-020-00550-8. Epub 2020 Sep 9. PMID 32902766
- [Background] Brkanovic S, Ivanisevic A, Miletic I, Mezdic D, Jukic Krmek S. Effect of Nano-Filled Protective Coating and Different pH Enviroment on Wear Resistance of New Glass Hybrid Restorative Material. Materials (Basel). 2021 Feb 5;14(4):755. doi: 10.3390/ma14040755. PMID 33562810